CLINICAL TRIAL: NCT04512027
Title: Effect of Prolectin-M; a (1-6)-Alpha-D-Mannopyranose on SarsCoV2 Viral Copy Numbers: A Proof of Concept, Open Label Randomized Controlled Trial
Brief Title: Prolectin-M in COVID-19 Patients Having Mild to Moderate Symptoms Not Requiring Oxygen Support.
Acronym: Prolectin-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Composite Interceptive Med Science (Industry)
Collaborators: Bioxytran Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIMED - 002- 2020
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
Keywords: ddPCR,; SarsCoV2 Copies
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolectin-M; a (1-6)-alpha-D-Mannopyranose class+Stand of care (Experimental): Tablet chewed for 5 days along and given alongside standard of care
  Interventions: Other: Prolectin-M; a (1-6)-alpha-D-Mannopyranose class; Other: Standard of Care
- Standard of Care (No Intervention): All patients will receive currently practiced standard of care medicines

INTERVENTIONS:
Other: Prolectin-M; a (1-6)-alpha-D-Mannopyranose class — A treatment to decrease viral load, detected through digital droplet PCR, in mild to moderate cases of RT-PCR positive COVID-19
  Arms: Prolectin-M; a (1-6)-alpha-D-Mannopyranose class+Stand of care
Other: Standard of Care — Currently approved standard of care for patients without symptoms requiring hospitalisation will be provided to all.
  Arms: Prolectin-M; a (1-6)-alpha-D-Mannopyranose class+Stand of care

SUMMARY:
A randomised controlled trial of open label Prolectin-M; a (1-6)-alpha-D-Mannopyranose among patients with RT PCR positive COVID-19 patients.

DETAILED DESCRIPTION:
SarsCoV2 has infected over 20 million people worldwide. The virus has a unique protein structure enabling it to rapidly infect and spread among the population. COVID19 is a global health emergency and has affected lives of all people irrespective of being infected. There are no proven therapies and a vaccine is yet to be approved for wide public usage.

Our study aims to test a hypothesis of physically blocking the spike protein from infecting the human cells, thus promoting its rapid excretion from the infected person.

We will randomise 10 subjects in this proof of concept trial and test the hypothesis by measuring the effect of Prolectin-M; a (1-6)-alpha-D-Mannopyranose in reducing the viral copy numbers over 5 days of treatment. The absolute copy numbers will be measured on digital droplet PCR developed by BioRad. A fall in copy numbers by 2-fold from baseline will be considered a positive treatment effect in this population. All standard care measures currently being practiced for these patients will be continued.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic and laboratory-confirmed diagnosis of COVID-19.
* Age ≥18 years and ≤45 years, male and non-pregnant female
* Identified within 72 hours of testing positive on RT PCR.
* Able to give informed consent to stay in institutional care and undergo 3 times collection of throat and nasal swabs over 7-day period; Day 1, Day 3 and Day 5 since randomization.

Exclusion Criteria:

* Oxygen saturation at admission ≤96%.
* High temperature ≥100 deg F (≥37.5 deg C) not controlled on oral doses of acetaminophen.
* Known history of diabetes on oral medications or insulin.
* IL-6 levels ≥ 3times of laboratory reference range and / or significantly elevated levels of CRP, serum ferritin or d-dimer.
* Lymphocyte / monocyte ratio ≤3 or neutrophil / lymphocyte ratio ≥5 or platelet count ≤150,000 cells per microliter
* On any chronic medications for more than 4 weeks before randomization or active malignancy or having any co-morbidity that increases risk of rapid disease progression.
* Previously tested positive and recovered from COVID-19

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-09-19 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
SarsCoV2 viral copy number | 7 days from randomisation
  Change in absolute viral copy number

SECONDARY OUTCOMES:
b. Disease progression will be measured on a 7-point scale at 28 days. A 2-point change will be considered disease progression. | 28 days from randomisation
  7-point severity score (ordinal scale):
  1. Not hospitalized, no limitations on activities
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen;
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO);
  7. Death

CONTACTS AND LOCATIONS:
Locations (1):
- Mazumdar Shaw Medical Centre, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suo T, Liu X, Feng J, Guo M, Hu W, Guo D, Ullah H, Yang Y, Zhang Q, Wang X, Sajid M, Huang Z, Deng L, Chen T, Liu F, Xu K, Liu Y, Zhang Q, Liu Y, Xiong Y, Chen G, Lan K, Chen Y. ddPCR: a more accurate tool for SARS-CoV-2 detection in low viral load specimens. Emerg Microbes Infect. 2020 Dec;9(1):1259-1268. doi: 10.1080/22221751.2020.1772678. PMID 32438868
- [Background] http://medrxiv.org/lookup/doi/10.1101/2020.02.29.20029439